CLINICAL TRIAL: NCT02018497
Title: Essential Arterial Hypotension and Allostasis Registry
Brief Title: Essential Hypotension and Allostasis Registry
Acronym: ESSENTIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Luis Eduardo Medina, Researcher, CES University
Other Study IDs: LEMD001
Record Dates: First submitted 2013-11-29; First posted 2013-12-23 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Blood Pressure; Depression; Panic Attack; Fibromyalgia; POTS; Inappropriate Sinus Tachycardia; Coronary Heart Disease; Acute Coronary Syndrome (ACS); Acute Myocardial Infarction (AMI); Cerebrovascular Disease (CVD); Transient Ischemic Attack (TIA); Atrial Fibrillation; Diabetes Mellitus; Cancer; Systolic Heart Failure; Diastolic Heart Failure; Chronic Fatigue Syndrome; Syncope; Vasovagal Syncope
Keywords: Essential arterial hypotension; Arterial hypotension; Low blood pressure; Hypotension; Essential arterial hypertension; Syncope; Dysautonomia; Stress; Adaptability; Reactivity; Homeostasis; Allostasis; Allostatic load; Distress; Epigenetic; Plasticity
MeSH Terms: conditions — Depression; Panic Disorder; Fibromyalgia; Coronary Disease; Acute Coronary Syndrome; Cerebrovascular Disorders; Ischemic Attack, Transient; Atrial Fibrillation; Diabetes Mellitus; Neoplasms; Heart Failure, Systolic; Heart Failure, Diastolic; Fatigue Syndrome, Chronic; Syncope; Syncope, Vasovagal; Hypotension; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive patients who consult a cardiologist: Consecutive patients who consult a cardiologist - electrophysiologist since June 2006, regardless of the age or gender in the city of Medellin, Colombia. They could have consulted previously (considered as the enrollment date) if they had, at least, one measurement of their BP in supine position, and an immediate measurement of their BP in standing position that allows diagnosing their group of blood pressure. All patients have a record in paper and/or magnetic file and in OpenClinica.
  No interventions.

SUMMARY:
The essential arterial hypotension and allostasis registry is a prospective, observational research that has the purpose of demonstrating that essential blood pressure (BP) disorders and the associated comorbidities are a result of the inappropriate allostatic response to daily life stress. This required a functioning brain orchestrating the evaluation of the threat and choosing the response, this is a mind-mediated phenomenon. If the response is excessive it contributes to high BP, if deficient to low BP, and the BP itself will identify the allostatic pattern, which in turn will play an important role in the development of the comorbidities.

To do so, consecutive patients of any age and gender that visit a cardiologist's office in Medellin, Colombia, are recruited. Individuals are classified according to their arterial BP and allostasis and follow them in time to see what kind of diseases develops the most (including BP) in the follow up according to the categorization of the characteristic chosen and after adjustment for confounder's variables. In addition, stress events with their date are registered.

HYPOTHESIS

The causes of the diseases are multifactorial.

Physical, biochemical, psychological, social, and cultural dimensions of development dynamically interact to shape the health development process.

A person´s health depends on their:

1. Biological and physiologic systems
2. External and internal environment (a) physical, b) internal behavioural and arousal state as registered by the brain.
3. Their interaction.

The allostatic mechanisms to the internal and external stressors (allostatic load) involves a network composed by:

1. Functional systems; mediated by:

   1. The Autonomic Nervous System
   2. The endocrine system
   3. The immune system
2. Structural changes: whenever the internal and/or external stressors are long lasting and/or strength enough, they may induce changes in:

   1. Epigenetic, endophenotypes, polyphenism.
   2. Plasticity
3. The interaction between a) and b).

The network response do not affect exclusively the BP, propitiating the development of comorbidities, which may prompt strategies for prevention, recognition and ultimately, treatment.

The allostatic model defines health as a state of responsiveness.

The concept of psycho-biotype: The allostasis is the result of both: biological (allostasis) and psychological (psychostasis) abilities. It is proposed that both components behave in similar direction and magnitude.

Immune disorders may be associated with the development of cancer. High BP population has a higher sympathetic and lower vagal tone, this has been associated with a decrease in the immune´s system function.

Resources and energy depletion: Terms like weathering have been used to describe how exposures to different allostatic loads gradually scrape away at the protective coating that keeps people healthy. It is postulated that High BP individuals have more resources and energy.

DETAILED DESCRIPTION:
DEFINITIONS

ARTERIAL BLOOD PRESSURE CLASSIFICATION

Arterial Blood Pressure (ABP) is a complex physiological variable in regard to its measure, behavior between BP taken in the same visit at the office and between these and ABPM, chronobiology (different day time BP levels), evolution in time, meaning and classification.

Not appropriate approach or analysis may be addressed without taking into account all the BP characteristics that have demonstrated prognostic implications.

In order to arrive to the most comprehensive analysis, BP classification takes into account the following characteristics:

I. Cause of BP disorder

A. Primary or Essential: Not clear causes may be identified. Multiple mechanisms may be involved, obvious players and contributors, but no definitive cause.

B. Secondary: an identifiable cause is characterized.

.

II. The sitting, supine, standing BP and/or ABPM value

A. High arterial BP (HBP):

1. At the office: the average of the two systolic or diastolic sitting, supine, standing BP are considered.

   1. Office Supine SBP ≥140 mm Hg and/ or DPB ≥90 mmHg
   2. Diagnosis HBP: As single criteria in the abscence of ABPM
2. Ambulatory BP Monitoring (ABPM):

   1. 24 hrs: SBP ≥130; DBP ≥80 mmHg.
   2. Awake (06:00-22:00): SBP ≥135; DBP ≥85 mmHg.
   3. Night (22:00-06:00): SBP ≥125; DBP ≥70 mmHg.
3. Both at the office and ABPM always predominate ABPM:

   1. HBP in ABPM at 24 hrs, awake or night time, regardless of the office BP
   2. Masked hypertension (MHBP): HBP AWAKE in the ABPM and NBP or LBP at the office.

      B. Low BP (LBP) Since there are no clear limits in ABPM for LBP, only office supine SBP and/or DBP will be considered.

      SBP <90 DBP <60

      C. Normal BP (NBP) > 90 SBP <140 > 60 DBP <90 White Coat Hypertension (WCHBP): Normal BP AWAKE in the ABPM and HBP at the office.

      D. NIGHT BP
      1. Night HBP: HBP at night in the ABPM
      2. Night NBP: NBP at night in the ABPM
      3. Night LBP: LBP at nigth in the ABPM .

      III. The BP orthostatic response (Supine minus Standing [SUPINE] and Sitting minus Standing [SITTING], example: SUPINE OH, or SITTING OH)

      A. Orthostatic hypotension (OhypoT): Drop in BP upon standing
      * 20 mmHg if SBP is normal
      * 30 mmHg if SBP ≥140
      * 10 mmHg in DBP

      B. Orthostatic Hypertension (OhyperT) Rise in SBP upon standing ≥20 mmHg

      C. Orthostatic Normotension (ONT): No criteria for Ohypot or OhyperT

      .

      IV. The circadian component of BP

      A. Normal Dipper (NDBP): average decrease of SBP between day and night time greater than 10% and less than 20%

      B. Extreme Dippers (EDBP): greater than 20% fall

      C. Nondippers (NonDBP): less than 10% fall

      D. Reverse dippers (RDBP): night time BP higher than daytime average

      E. Abnormal early Morning BP Surge (BPS): A rise ≥50 mmHg.

      .

      V. BP response to treatment (requires office BP and ABPM)

      A. True Control HBP (TCHBP): NBP at the office and the ABPM AWAKE

      B. True Resistant HBP (TRHBP): HBP at the office and the ABPM AWAKE

      C. False Control HBP (FCHBP): NBP at the office and HBP in the ABPM AWAKE

      D. False Resistant HBP (FRHBP): HBP at the office and NBP in the ABPM AWAKE

      Patients must be in the absence of medication for Essential hypotension diagnosis and hypotension must be dismissed as a secondary manifestation of another disease or other condition such as dehydration, medication causing hypotension for other conditions or secondary dysautonomia.

      There are 3 types of orthostatic hypotension Initial: in the first 30 sec. after assuming the standing position Classic: It occurs between the 1st and 3rd min. Late: It occurs between 5 and 45 min. later (no patients within this category)

      ESTIMATION OF TARGET-ORGAN DAMAGE Electrocardiogram, Doppler color echocardiogram, creatinine and urinalysis, lipid and metabolic profile and microalbuminuria are requested to the patients; carotid Doppler is also requested in patients with suspect of disorder.

      ARTERIAL HYPERTENSION TREATMENT. The treatment starts with a low-sodium diet (by nutritionist whenever possible), increase in fruits and vegetables intake, weight loss, aerobic exercise, stop smoking, and changes in lifestyle.

      The pharmacological first step is the use of IECAs (ARA II if there is cough), calcium channel blockers, the use of diuretics like the Hydrochlorothiazide 12.5mg (or up to 25mg). If there is orthostatic hypotension, it is considered to start with Amlodipine. In those patients with tachyarrhythmia, heart failure or coronary disease Beta blockers are chosen. Alpha blockers are the last step therapy.

      ESSENTIAL HYPOTENSION TREATMENT The treatment starts with the use of non-pharmacological measures consisting of postural hygiene (avoid assuming the standing position abruptly, avoid staying in the standing position for too long), eat salty (10 g), drink more than 2 liters of water per day, do aerobic exercises, and raise the head of the bed. If there is not improvement, the patient can wear gradient tights up to the waist. Next step is start Fludrocortisone 0.05 daily or every other day. The last step is Midodrine (from 5 to 20mg daily, distributed at 06:00, 10:00 and 14:00 hrs or when needed, avoid it after 6:00 pm). Counterpressure maneuvers are recommended if there is a threat of syncope.

      ALLOSTASIS

      For the effects of what is mentioned here, allostasis is defined as the ability to maintain homeostasis through the neuroendocrine and immune response to the stress of any type. There is experimental evidence, measuring the sympathetic nerve activity during the mathematical stress with microneurography of the peroneal nerve (muscle sympathetic nerve activity or MSNA) that the response may be increasing, neutral or decreasing.

      The alterations in blood pressure are considered objective, which may be the result of strategies and different responses to stress (adaptability), through the neuroendocrine system (mainly the sympathetic nervous system).

      The following variables are evaluated to describe the Allostasis:

<!-- -->

1. SYMPTOMS OF HYPOTENSION: postural dizziness, dizziness after squatting, dizziness during childhood or adolescence (in elementary school, high school and occasionally in college) during the mass, at public events, religious processions or military parades. It is also taken into account the previous diagnosis of low pressure or "hypoglycemia" (which in our culture mainly refers to symptoms of orthostatic hypotension).
2. HISTORY OF NEURALLY MEDIATED SYNCOPE OR VASOVAGAL SYNCOPE diagnosed by the scores of Calgary or Tilt-test; or vasovagal syncope (syncope caused by seeing blood, a venipuncture or donating blood; pain, by seeing or speaking about dramatic things, when coughing, swallowing, defecating, urinating, laughing, or other situations). If these situations occur with significant dizziness or pre-syncope, but not syncope itself, it is called vasovagal component.
3. BLOOD PRESSURE: Low BP

The allostasis is classified as:

1. Hypo-allostasis: presence of at least one of the followings:

   1. Symptoms of hypotension and/or
   2. Neurally mediated syncope (clinical or at the tilt-test) or vasovagal syncope and/or
   3. Hypotension at the office or at the tilt-test
2. Normal-allostasis: normal blood pressure and no symptoms of hypotension, no neurally mediated syncope or vasovagal syncope (spontaneous or induced in the tilt table test) and no presence of hypotension. Include those who develop permanent hypertension after 65 yo. After this age, structural components mainly in the Windkessel vessels, may contribute more than the increased sympathetic tone to the hypertension phenomenon. For end points analysis, patients developing Hypertension after 65 yo are considered hypertensives in their BP group, but normal in the adaptability.
3. Hyper-allostasis: Arterial hypertension starting before 66 yo, with no identifiable cause, no symptoms of hypotension, no neurally mediated syncope or vasovagal syncope.

Allostasis scores (scores between 1 and 7 apply for hypo-allostasis only)

1. Only symptoms
2. Only essential hypotension
3. Only neurally mediated syncope
4. 1 and 2
5. 1 and 3
6. 2 and 3
7. 1, 2 and 3
8. Normotensive
9. Hypertensive
10. The patient does not remember

Thus then, 3 groups of blood pressure are recognized at the moment of evaluating their impact on the comorbidities:

1. Normotensive
2. Hypotensive
3. Hypertensive, that in turn can be:

   1. Hypertensive since the admission
   2. Previously hypotensive
   3. Previously normotensive

METHODS

Cohort.

LABORATORY EXAMINATIONS

Complete blood count Basal glycemia and 2 hr post-load 75 g glucose Insulinaemia Glycated hemoglobin Serum ferritin Thyroid stimulating hormone and sometimes free thyroxine Sodium and serum potassium Uric acid Lipid profile Creatinine Basal serum cortisol and/or post-Adrenocorticotropic hormone 24-hr urinary free cortisol Post-dexamethasone cortisol: in those with high cortisol with not recognized cause Microalbuminuria Others depending on the case, such as: 24-hr urine catecholamines (Epinephrine, Norepinephrine and Metanephrines), gliadin antibodies, vanillylmandelic acid, parathyroid hormone, vitamin B12, folic acid, ANAs, testosterone, creatinine clearance, antibodies against human hemoglobin in stool, hypersensitive reactive C protein, 24-hrs urinary sodium, brain natriuretic peptide, etc.

There is not a single laboratory to make the blood tests, so there are different values of normality for some tests.

PHYSICAL EXAMINATION

ANTHROPOMETRIC MEASUREMENTS:

In every medical consultation, the patient is weighed wearing trousers or skirt. The waist is measured at an equidistant level between the last rib and the iliac crest. The hip is measured at the level of the greater trochanter. Finally, the size that appears in the identity card of the patient, or the latest measurement is written down. After May 2016 measurements are taken in the office.

TAKING OF BLOOD PRESSURE:

It is performed using a mercury sphygmomanometer from Tycos brand (it is revised annually in accordance with the current rules of the Ministry of Health), and it is controlled that the mercury column falls to 2 mm per second.

The bracelet must cover approximately the 80% of the forearm. We have three sizes of bracelets as needed, including a pediatric bracelet. This should be positioned at heart level.

The appearance of the first sound and the disappearance of Korotkoff sounds are taken as systolic and diastolic BP respectively.

About 6 BP measurements are taken, two on supine position and the second one after 5 min. supine, this second supine value is the one used to calculate the BP drop upon standing. Later, and having the bracelet previously inflated, the BP is taken immediately once the up-right position is assumed (first 30 sec). Then, additional pressures are taken at the first, second and third min.

Since November the 30th, 2017, two additional BPs will be taken in a seated position; these will be taken at the beginning of the BP taking session. The patient will be seated comfortably with their right arm resting at the heart level. The BPs, HRs, COs and SVRs will be taken first after one minute of having the patient sit comfortably and then again after two minutes. Later on, the patient will assume the first supine position and the protocol continues as explained previously; however, the interval between the two BPs taken at the supine position will be of one and three minutes.

Starting on January 2018, an immediate standing BP after seated position will be taking.

Invasive beat to beat BP taken was no longer used since March 2020 because the COVID-19 Pandemic. Few patients have been seen since then, BP is taken with mercury sphygmomanometer always in sitting position and sometimes, in supine and standing position.

The same process is fulfilled for the HR, taken in 15 sec. During the taking of blood pressure neither the patient nor the doctor talk, and it is avoided making any comments that might alter the patient psychologically, and potentially modify their BP levels. The patient is asked to have an empty bladder and the Physician tries to support the patient´s arm at the heart level in every position.

NON-INVASIVE BEAT TO BEAT BP MONITORING Non-invasive, beat to beat, BP monitoring and Cardiac Output (CO) and Systemic Vascular Resistance (SVR) started to be used since May 2017 to measure BP, HR, CO, SVR. CNAP Monitor 500, CNSystems, is CE and FDA approved. It is intended to be use in every consecutive patient.

Instructions:

1. Rings, bracelets, and wristwatches should be withdrawn from the right arm.
2. Fingers in the cuffs should not be bending since this could increase BP artificially.
3. The arm will rest beside the body, relaxed.
4. When standing, the physician or person taking BP should take the patient´s right arm and help him stand up in an attempt to decrease the arm´s movement and avoid interference on the recording.
5. The forearm is kept at the heart level.
6. A screen´s photography will be taken with the cellphone after every BP measure (8).
7. A label is placed on the recording just after the seating position and before standing.
8. If the immediate standing BP taken shows a drop in the BP but systemic vascular resistance (SVR) and cardiac output (CO) are those of the supine position then the BP won´t be registered and a picture should be taken immediately SVR and CO are recalculated.
9. If BP starts to rise, review that fingers in the cuff are straight.
10. If in doubt, make a manual measure of the BP.
11. BP and HR date along with SVR and CO will be introduced in the fields of the BP and HR taken with the sphygmomanometer and usual physical examination. New fields were created for SVR and CO.
12. The completed data is introduced as 3 attachment files for further analysis.

ELECTROCARDIOGRAM (HEWLETT PACKARD AND MORTARA) A careful reading of each plot is made in which the HR, PR and cQT intervals, and QRS complex are recorded (automatic measurements).

24 HOURS ECG MONITORING (HOLTER) It is specified the patient rhythm, if is under medication that may affect the heart rate variability (HRV) and, it is recorded the name and type of drug. The number of supraventricular and ventricular premature complexes are counted.

The components of heart rate variability (HRV) allows calculating the sympathovagal balance (SVB) in 24 hrs, in the day (06:00 to 22:00) and at night (22:00 to 6:00).

Low frequency (LF), high frequency (HF), very low frequency (VLF), Total power (TP) LF or HF one = LF or HF x 100/ TP-VLF SVB = LFone/HFone

AMBULATORY BLOOD PRESSURE MONITORING (ABPM) The systolic and diastolic BP and HR are registered in 24 hrs, in the day and at night, as in the 24-hr Holter monitoring. This test is requested for all patients in order to define the presence of white coat hypertension or masked hypertension and to define an effective treatment.

Morning surge in SBP: It results from the difference between the averages of SBP taken in the first 2 hrs from awakening and the lower nighttime.

COLOR DOPPLER ECHOCARDIOGRAM AND/OR STRESS ECHOCARDIOGRAM It is made the measurement of the heart and if the response to stress is positive or negative.

The ejection fraction (EF) is usually measured by the technique of Simpson or in a qualitative way.

Body surface area = (weight x height / 36) X 1/2 Cardiac mass = 1.05 [(LVDD + SW + PW)3 - LVDD3] - 14 Cardiac mass index = cardiac mass / body surface area

ABDOMINAL ULTRASOUND It is recorded the presence of fatty liver and abdominal aortic aneurysm

UPPER GASTROINTESTINAL ENDOSCOPY AND COLONOSCOPY The main findings are recorded

CORONARY ANGIOGRAPHY Indication: For those who belong to the protocol and will indicate it, it is tried that the indication belongs to a score between 7 and 9 (appropriate test for a specific indication) of the recommendation of the working group aforementioned.

1. In patients with symptoms of acute coronary syndrome or positive test for myocardial ischemia in individuals with moderate or high cardiovascular risk
2. In patients with sustained ventricular tachyarrhythmias with unidentifiable cause that stop spontaneously or require resuscitation
3. In patients with left ventricular dysfunction at basal conditions (ejection fraction <40%) and evidence of viability in the affected segments.
4. Evidence of new segmental alteration of motility of unknown etiology.
5. Suspected ischemic mitral regurgitation or interventricular septal defect.
6. Presence on the CT scan of lesions >50% on the left main trunk or other vessels, or possibly obstructive lesions of debatable severity in symptomatic patients (when in the left main trunk, also in asymptomatic patients)

It is classified according to the obstruction to coronary flow as follows:

* Lesion <50%, non-obstructive (if not the left main trunk)
* Between 50-69%, intermediate lesion (if not the left main trunk)
* >70% or >50% of the left main trunk, it is a significant obstructive lesion. It is neither specified the number of affected vessels nor the vessel diameter.

ELECTROPHYSIOLOGICAL STUDY The patient must be in a fasting state and stop taking medications that affect the study for at least 5 half-lives. It is made by puncturing the right femoral vein, electro-catheters are placed in the high right atrium, in the bundle of His and in the right ventricular apex. It is stimulated the double of the thresholds to 3 cycle lengths (600, 500 and 430 ms) and three extra cycles, starting at 350 ms, and with successive decreases of 10 ms until the refractory period is found.

The study is made at basal conditions and in presence of Isoproterenol up to 4 micrograms/min; the sedation is obtained with Midazolam, administered 10 min. before starting the measurements.

Sinus function tests: Sinoatrial conduction time (by Narula method), the sinus node recovery time (SNRT) and the corrected sinus node recovery time (CSNRT)). For the SNRT, it is stimulated to several cycle lengths for one min, with decreases of 100 ms up to 430 ms, and the longest pause is considered as the recovery time; if greater than 1500 ms is considered abnormal.

The CSNRT is the result of SNRT minus the cycle length of the patient. It is considered abnormal 500 ms or more (sensitivity of 85% and specificity of 90%). Additionally, at five min, it is evaluated the response of the HR to the infusion of 3 micrograms of Isoproterenol per min. (an increase of 25% from basal HR) and the intrinsic HR.

This latter is made by administering Atropine 0.04 mg/kg and propranolol 0.2 mg/kg, the intrinsic HR is dependent on the age, and is calculated as follows:

118.1 - (0.57 x age), for people under the age of 45 the value is adjusted +14% and for people over the age of 45 +18%.

Indication:

1. In patients with syncope and ischemic heart disease, when the initial evaluation suggests an arrhythmic cause.
2. In patients with syncope and bundle branch block, when the noninvasive evaluation has not clarified the diagnosis.
3. When brief and sudden palpitations precede syncope, when the noninvasive evaluation has not clarified the diagnosis.
4. In some cases of Brugada syndrome, arrhythmogenic right ventricular cardiomyopathy and hypertrophic cardiomyopathy.
5. In high-risk patients in whom other methods have not clarified the diagnosis.

TILT TABLE TEST The patient is connected to the noninvasive BP beat to beat monitor. (Task Force Monitor).

The patient must be fasting for at least 4 hrs; should stay 5 min. in supine position and then is tilted at 60 degrees for 20 min. Then, it is administered 400 micrograms of sublingual nitroglycerin for 20 min. more. The tilt table test (TTT) is considered positive if the patient presents syncope or if the systolic blood pressure is lower than 60 mmHg. The hemodynamic variables, the HR variability, and the BP are written down for those patients who have these values available.

Other diagnoses written down on the TTT are:

* Postural orthostatic tachycardia syndrome (POTS):
* Inappropriate sinus tachycardia (IST): It is defined as a HR greater than 90 bpm in supine position.
* Orthostatic hypotension (OH):

Fall in the systolic BP ≥20 mmHg or in diastolic BP ≥10 mmHg, at any time of the TTT.

. Orthostatic Hypertension: rise in SBP ≥20 mmHg.

* Asystole: Isoelectric line that last for more than 3 sec. on the electrocardiogram plot. The duration in sec. of the asystole is recorded.
* Chronotropic incompetence (CI):

It refers to the inability of the heart to increase the HR more than 10% when standing up within the first 10 min, and if the HR in supine <70 bpm. Also, if this criterion is not met but the HR to 60 degrees is lower than 65 bpm.

Indication:

Single syncope episode of unknown origin in high risk patients, or recurrent syncope in absence of organic heart disease; or in presence of organic heart disease if cardiac etiology was previously dismissed.

To show to the patient that he/she has this mechanism of syncope. To discriminate between reflex and orthostatic syncope To differentiate syncope from epilepsy To diagnose patients with recurrent unexpected falls To evaluate patients with recurrent syncope and psychiatric disease Many patients referred by other colleagues already have the TTT.

CAROTID SINUS MASSAGE (CSM) It is made during the TTT

Contraindications for the accomplishment of the procedure:

1. History of cerebrovascular disease
2. Acute myocardial infarction in the previous 3 months, or
3. Presence of carotid bruit during the neck auscultation. The test consists of doing pressure and circular movements during 10 sec. on each carotid sinus, allowing an interval of 1 min. between both sides. The massage is made at 0 and 60 degrees tilt. It is considered a vasodilatory response if the systolic BP falls at least 50 mmHg, and chronotropic response if an asystole last 3 or more sec. If this latter occurs, it is expected the patient to recover and the carotid massage is repeated after applying atropine 1 mg. If still positive for syncope it is considered a mixed response to the CSM.

OTHER EXAMINATIONS These tests are requested as needed to clarify other findings. 1. Computerized axial tomography of brain, heart 2. Brain or heart nuclear magnetic resonance 3. Polysomnography 4. Meta-iodo-benzyl-guanidine 5. Carotid, renal and lower limbs arterial Duplex 6. Heart or other structures biopsy 7. Others

DATABASE We have over 1100 variables in OpenClinica 3.13

UPDATING INFORMATION It is made through the consultations, phone calls or emails sent to the patient email address. The patients should be contacted annually if possible.

Requested information:

1. Updating of telephone number, cell phone number and e-mail addresses
2. Full treatment
3. Patient is questioned about new family histories
4. Patient is questioned about new comorbidities, when were they diagnosed and by whom, following the existing comorbidities in the database.
5. Patient´s current weight and exercise
6. Paraclinical laboratory tests.

COMORBIDITIES DIAGNOSTIC CRITERIA

1. Depression:

   The diagnosis is made by a psychiatrist and/or if the patient meets the criteria of DSM IV. If there is difference between the psychiatric diagnosis and the DSM IV criteria, the diagnosis made by the psychiatrist prevails.
2. Panic attack:

   The diagnosis is made by a psychiatrist, the DSM IV criteria or both, the diagnosis made by the psychiatrist prevails.
3. Fibromyalgia:

   It is diagnosed by a rheumatologist.
4. Postural Orthostatic Tachycardia Syndrome (POTS), not associated with hypotension.:

   * Increase in the HR >30 bpm when standing up.
   * Increase in the HR >40 bpm when standing up, between 12 and 18 years old.
   * HR >120 bpm during the first 10 min. of standing up
5. Inappropriate sinus tachycardia:

   It is the HR average during the 24-hr Holter monitoring >90 bpm, in absence of secondary cause.
6. Coronary heart disease:

   It is diagnosed by the ACS criteria or by the abnormal coronary angiogram.
7. Acute coronary syndrome (ACS):

   It refers to clinical, enzymatic, electrocardiographic, echocardiographic or angiographic findings, diagnosis of acute coronary disease. It should be dismissed the cocaine abuse, Prinzmetal's angina and Takotsubo cardiomyopathy. This latter is classified as such in a separate box.
8. Acute myocardial infarction (AMI):

   Term used when there is evidence of myocardial tissue necrosis in the clinical spectrum of myocardial ischemia.

   Ischemic symptoms. New changes or presumed new in the ST segment and T wave, or a new LBBB. Development of new Q waves on the ECG Evidence by images of loss of viable myocardium, or the emergence of a segmental defect in the motility.

   Identification of an intracoronary thrombus in an angiography or autopsy.

   Criteria for prior myocardial infarction:

   Pathological Q waves on the ECG, with or without symptoms, in absence of non-ischemic causes.

   Evidence by images of loss of viable myocardium, which is thinner and does not contract, in absence of non-ischemic cause.

   Pathological findings of a previous MI.
9. Cerebrovascular disease (CVD) or transient cerebral ischemia (TCI):

The TCI has traditionally been considered as a deficit lower than 24 hrs in duration, and so it is considered in this protocol. Well-founded evidence suggests duration lower than 60 min, and no evidence of nerve damage proved by CT scan or MRI.

10. Atrial fibrillation: Baseline low amplitude oscillations with irregular rhythm on the ECG or at Holter monitoring (30 sec)

11. Diabetes mellitus: Fasting glucose > 126 mgs/dl Occasional glucose > 200 mgs/dl with symptoms Glucose load (75 g): > 200 at 2 hrs A1C > 6.5.

12. Cancer: It is diagnosed by an oncologist.

13. Systolic or diastolic heart failure: Patients should be symptomatic. It is considered systolic if the ejection fraction is decreased, otherwise, it is considered diastolic. In case of being diastolic, it should be dismissed other causes of dyspnea, such as lung diseases.

14. Chronic fatigue syndrome or idiopathic chronic fatigue: Persistent or chronic fatigue, clinically evaluated, unexplained, which lasts for 6 or more consecutive months, of recent onset, not explained by exercising, not improved substantially with rest and that produces a substantial reduction in previous levels of occupational, social, educational and personal activities.

The patient must have 4 of the following symptoms, which must have persisted or be recurrent for 6 or more consecutive months of illness, and must have not been preceded by fatigue: a) self-reporting of poor short-term memory or decreased ability to concentrate, as severe as to alter the previous functional ability, b) dry throat, c) armpit and cervical adenopathies, d) muscle pain, joint pain without redness, deformity or swelling, de-novo headache, e) unrefreshing sleep, and malaise post exercise that lasts more than 24 hrs.

15. Syncope: It refers to the transient loss of consciousness secondary to cerebral hypoperfusion, characterized by sudden onset, short duration, and spontaneous and complete recovery.

16. Vasovagal syncope Emotion mediated syncope or orthostatic stress, usually preceded by autonomic activation prodromes (diaphoresis, pallor, nausea). It includes situational syncope and carotid sinus hypersensitivity.

PSYCHO BIOTYPE EVALUATION

Design to study in depth the Psycho Biotype hypothesis. It consist of consecutive patients of each BP group to whom the following test are apply:

1. Big Five Questionary (BFQ) for personality.
2. Modified Coping Scale (Scale of modified coping strategies)
3. Zung questionary for depression and anxiety
4. MINI in those patients with moderate or severe depression and/or anxiety at the Zung questionary, apply by a psychiatrist

GENERAL OBJECTIVE To demonstrate if the essential arterial BP group and/or the adaptability are clinically important and try to identify the mechanism involve.

SPECIFIC OBJECTIVES To demonstrate that the three groups of blood pressure differ in the numbers taken as much in the doctor's office as in the ambulatory BP monitoring.

To inquire what variables are different between the groups of BP. To inquire which comorbidities are more associated with each group of blood pressure and evaluate whether the differences persist after a multivariate analysis. The same will be done with the adaptability groups.

To provide hypotheses or evidences to explain the findings of the study.

DESIGN OF THE STUDY This is an observational, analytic, cohort type study that aims to compare the differences between groups of patients classified according to their BP numbers and their adaptability.

To this end, variables of the clinical, paraclinical, imaging and comorbidities profile will be evaluated.

The database is designed to be flexible. It allows choosing different conditions in different variables. The diagnoses have 3 options: No, New and Old. It is recorded the date of the physical examinations, the diagnoses and the paraclinical results to ensure accuracy in the calculation of the age and the relationship between the different variables during the analysis.

The reports will be of prevalence (cross-sectional) and incidence (cohort). To evaluate the significance between the groups of blood pressure depending on morbidities and other variables, it is used a generalized linear model by adjusting the effect of the response variable based on the age, gender and tension group in all cases. In some cases, and when the response variable requires it, it is added the body mass index (BMI). When the response variable is qualitative, it is used a logit link function and it is obtained the corresponding Odds ratio with confidence intervals to 95%; while if the variable is quantitative it is used the identity function. Finally, the multiple comparison test of Tukey-Kramer is made in order to compare the groups of tension with a significance level of 0.05.

To evaluate the relationship between the blood pressure groups and the comorbidities, and other variables, the free events survival rates among participants using a Kaplan Meir survival curves, adjusted for age and other related variables.

For the diagnosis of coronary disease, it was used a generalized linear model in which was evaluated the adjustment of the effect in the groups of tension by age, gender, and body mass index (BMI), diabetes mellitus (DM), systolic and diastolic blood pressure in supine, total cholesterol, HDL cholesterol, smoking, and blood pressure group. Variables were selected by the method of Backward maintaining in the model those variables with a significance level of 0.05.

LIMITATIONS:

1. Because patients were recruited at the doctor's office, some of them may decide not to take the required tests or decide not to come back.
2. Some insurance companies may not provide some test, like the Ambulatory blood pressure monitoring.
3. The attending practitioner may be busy with too much work and has not available time to see the patients opportunely.
4. The blood tests can be done at different sites and by different operators.
5. Black population is not represented in this sample.

ELIGIBILITY:
Inclusion Criteria:

* Any patient regardless of the age of gender

Exclusion Criteria:

* Any non-correctable secondary cause of increase or decrease in blood pressure
* or a pathology that alters the prognosis before the entrance of the patient into this registry.
* nephropathy prior to the admission,
* familial dyslipidemia,
* previous gastric bypass,
* pre-existing heart failure,
* chemotherapy-induced cardiotoxicity,
* arrhythmogenic right ventricular dysplasia,
* long QT syndrome,
* hypertrophic cardiomyopathy
* restrictive cardiomyopathy or sudden death syndromes other than coronary disease
* Down syndrome,
* having one single kidney before entering to this registry,
* polycystic kidney,
* disability to continue with the treatment
* organ transplantation (other than cornea),
* HIV positive,
* homocystinuria,
* myelomeningocele,
* autoimmune diseases,
* paraplegia,
* chronic infections (TB),
* myocarditis of any cause,
* blood dyscrasia with coagulation disorders,
* history of pulmonary embolism,
* sustained or non-sustained ventricular tachycardia,
* idiopathic tachycardia associated with syncope which is not cured by radiofrequency ablation,
* pulmonary hypertension,
* diabetes insipidus,
* COPD,
* Gitelman syndrome,
* Cervical cancer associated with human Papillomavirus,
* multiple sclerosis,
* hemochromatosis,
* not compact ventricle.

It is important to emphasize that all of these patients, currently excluded from the registry, may be studied in the future, they keep on follow-up and taken 6 BP.

Additionally it is planned to compare the evolution of patients with secondary causes of hypertension or hypotension with essential disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients that visits a cardiologist's office in Medellin, Colombia. The population consists of patients of any age and gender, which are classified according to their blood pressure in: normotensive, hypertensive and hypotensive, they are also classified according to their adaptability in hypo, normo and hyper.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1995-01; Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between Blood pressure group and comorbidities | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Comorbidities: As describe in the protocol, as a summary: 1) cardiovascular, 2) metabolic, 3) Endocrine, 4) psychiatric disorders: depression and panic disorder, 5) orthostatic intolerance: neurally mediated syncope, vasovagal syncope, inappropriate sinus tachycardia, Postural orthostatic syndrome, carotid sinus hypersensitivity; 6) others: chronic fatigue syndrome, fibromyalgia, arthritis, autoimmune diseases, pulmonary thromboembolism, OSA (obstructive sleep apnea), Alzheimer disease, Parkinson disease, others dementias, epilepsia, nephropathies, and others.
  Cardiovascular mortality Total mortality
Relationship between adaptability group and comorbidities | A 7-year prospective study
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable. Comorbidities: As describe in the protocol, as a summary: 1) cardiovascular, 2) metabolic, 3) Endocrine, 4) psychiatric disorders: depression and panic disorder, 5) orthostatic intolerance: neurally mediated syncope, vasovagal syncope, inappropriate sinus tachycardia, Postural orthostatic syndrome, carotid sinus hypersensitivity; 6) others: chronic fatigue syndrome, fibromyalgia, arthritis, autoimmune diseases, pulmonary thromboembolism, OSA (obstructive sleep apnea), Alzheimer disease, Parkinson disease, others dementias, epilepsia, nephropathies, and others.
  Cardiovascular mortality Total mortality
Relationship between blood pressure group, adaptability group and comorbidities | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable. Comorbidities: As describe in the protocol, as a summary: 1) cardiovascular, 2) metabolic, 3) Endocrine, 4) psychiatric disorders: depression and panic disorder, 5) orthostatic intolerance: neurally mediated syncope, vasovagal syncope, inappropriate sinus tachycardia, Postural orthostatic syndrome, carotid sinus hypersensitivity; 6) others: chronic fatigue syndrome, fibromyalgia, arthritis, autoimmune diseases, pulmonary thromboembolism, OSA (obstructive sleep apnea), Alzheimer disease, Parkinson disease, others dementias, epilepsia, nephropathies, and others.
  Cardiovascular mortality Total mortality

SECONDARY OUTCOMES:
Relationship between blood pressure group, habits and anthropometric, metabolic, endocrine, Electrocardiogram, Holter, ambulatory blood pressure monitoring (ABPM) | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Habits: smoke and drink
  Anthropometric variables: Body mass index, waist, hip
  Metabolic variables: Fasting glucose, 2 hs postprandial plasma glucose, insulin plasma levels, homoeostasis model assessment (HOMA), total cholesterol, LDL, HDL, triglycerides.
  Endocrine variables: plasma cortisol, free cortisol in 24 hs. urine, epinephrine, norepinephrine, metanephrines, vanilmandelic acid, ACTH, aldosterone, renin, thyrotropine, free thyroxine, triiodothyronine, testosterone
  Electrocardiogram: HR; PR interval, QRS complex, cQT interval
  Holter variables: HR, standard deviation of NN intervals (SDNN) and sympathovagal balance, at day, night and 24 hs.
  ABPM: Systolic, diastolic, and heart rate, at day, night and 24 hs., BP matinal surge.
Relationship between blood pressure group, adaptability group, habits anthropometric, metabolic, endocrine, electrocardiographic, Holter, ambulatory arterial blood pressure monitoring. | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable.
  Habits: smoke and drink
  Anthropometric variables: Body mass index, waist, hip
  Metabolic variables: Fasting glucose, 2 hs postprandial plasma glucose, insulin plasma levels, HOMA, total cholesterol, LDL, HDL, triglycerides.
  Endocrine variables: plasma cortisol, free cortisol in 24 hs. urine, epinephrine, norepinephrine, metanephrines, vanilmandelic acid, ACTH, aldosterone, renin, thyrotropine, free thyroxine, triiodothyronine, testosterone
  Electrocardiogram: PR interval, QRS complex, Heart rate, cQT interval
  Holter variables: HR, SDNN and sympathovagal balance, at day, night and 24 hs.
  ABPM: Systolic, diastolic, and heart rate, at day, night and 24 hs., BP matinal surge.
For metabolic disorders what it matters the most: the anthropometric variables vs blood pressure group vs adaptability group | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Adaptability group: 1) Hyper adaptable, 2) normal adaptability and 3) hypo adaptable.
  Habits: smoke and drink, exercise
  Anthropometric variables: Body mass index, waist, hip
  Metabolic and other variables: Fasting glucose, 2 hs postprandial plasma glucose, insulin plasma levels, HOMA, total cholesterol, LDL, HDL, triglycerides; thyrotropine,
  Holter variables: HR, standard deviation of NN intervals (SDNN) and sympathovagal balance, at day, night and 24 hs.
  ABPM: Systolic, diastolic, and heart rate, at day, night and 24 hs., BP matinal surge.
Relationship between adaptability group, habits and anthropometric, metabolic, endocrine, Electrocardiogram, Holter, ambulatory blood pressure monitoring (ABPM) | A 7-year prospective study
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable.
  Habits: smoke and drink Anthropometric variables: Body mass index, waist, hip
  Metabolic variables: Fasting glucose, 2 hs postprandial plasma glucose, insulin plasma levels, HOMA, total cholesterol, LDL, HDL, triglycerides.
  Endocrine variables: plasma cortisol, free cortisol in 24 hs. urine, epinephrine, norepinephrine, metanephrines, vanilmandelic acid, ACTH, aldosterone, renin, thyrotropine, free thyroxine, triiodothyronine, testosterone
  Electrocardiogram: PR interval, QRS complex, Heart rate, cQT interval
  Holter variables: HR, SDNN and sympathovagal balance, at day, night and 24 hs.
  ABPM: Systolic, diastolic, and heart rate, at day, night and 24 hs., BP matinal surge.

OTHER OUTCOMES:
Syncope Registry | Up 100 weeks
  Clinical syncope characteristics (age of first syncope, number of syncope episodes, trauma, duration, clinical score, convulse, sphincter relaxation, etc.) Syncope cause Blood pressure group Adaptability group Prognosis
Tilt table testing (TTT) registry | Up to 100 weeks
  TTT protocol: describe the protocol, the time at positive response, nitroglycerine use, autonomic and hemodynamic variables.
  TTT outcome for syncope: positive or negative TTT other outcomes: 1) Chronotropic incompetence, 2) arterial orthostatic hypotension, 3) carotid hypersensitivity, 4) POTS, 5) IST The relationship between TTT results and Clinical score for syncope in regard to: syncope behaviour and other orthostatic intolerance entities, symptoms and comorbidities.
  The relationship between neurally mediated syncope response at the TTT and comorbidities.
Sinus node function at the electrophysiological study (EPS) | Up to 100 weeks
  EPS variables: AH, AV, CL, sino atrial conduction time (SACT), sinus node recovery time (SNRT), corrected sinus node recovery time (CSNRT), response to Isoproterenol, intrinsic heart rate Diagnosis: control, sick sinus syndrome, IST, chronotropic incompetence at the TTT HR at the ECG HR at the Holter monitoring HR at the TTT HRV at the Holter monitoring Syncope, cardiac or neurally mediated HR at the physical treadmill test Relationship with the blood pressure group Relationship with the adaptability group
Score for coronary artery disease | Up to 200 weeks
  Define how the blood pressure group and/or the adaptability group may add to the already known and include in this registry, in the diagnosis of cardiovascular complications as coronary artery disease, cerebrovascular disease, peripheral artery disease, nephropathy.
Neurally Mediated Syncope: further of the transient lost of consciousness (TLC) | A 7-year prospective study
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable. Comorbidities: As describe in the protocol, as a summary: 1) cardiovascular, 2) metabolic, 3) Endocrine, 4) psychiatric disorders: depression and panic disorder, 5) orthostatic intolerance: neurally mediated syncope, vasovagal syncope, inappropriate sinus tachycardia, Postural orthostatic syndrome, carotid sinus hypersensitivity; 6) others: chronic fatigue syndrome, fibromyalgia, arthritis, autoimmune diseases, pulmonary thromboembolism, OSA (obstructive sleep apnea), Alzheimer disease, Parkinson disease, others dementias, epilepsia, nephropathies, COPD, and others.
  Mortality
Psychobiotype: relationship between biological and psychological variables | Up to 100 weeks
  Blood pressure group: 1) Essential arterial hypotension, 2) normotension and 3) Essential arterial hypertension.
  Adaptability group: Hyper adaptable, normal adaptability, hypo adaptable.
  Psychiatric variables:
  1. Big Five Questionary (BFQ) for personality.
  2. Modify of the Coping Scale (Scale of modified coping strategies)
  3. Zung questionary for depression and anxiety
  4. MINI in those patients with moderate or severe depression and/or anxiety at the Zung questionary
The role of high sodium intake in the development of essential hypertension. Comparison between essential hypotension (high sodium intake) vs normotension population (normal or low sodium intake) in the follow-up. | 4 years
  High sodium intake in the diet is recognized as a risk factor for hypertension development.
  Essential hypotension population is advised to increase the sodium (at least 10 grams a day) and water intake (at least 2 liters a day), or as much as possible, several have taken Fludrocortisone (is not a exclusion criteria). Normal blood pressure population are advised to have a normal or low sodium intake. Physical exercise is recommended in both groups.
  This registry is a good opportunity to test how important sodium diet is to induce hypertension, or if by the contrary adaptability could prevail over high sodium intake in this registry.
  Blood pressure groups: essential hypotension and normotension and those with new essential hypertension. Adaptability groups.
  The results will be adjusted for age, gender and BMI.
White coat effect in the heart rate or masked bradycardia. | 1 year
  Consistent bradycardia in the ECG at the office and normal HR in the holter monitoring or the contrary.
  There are patients with complaints that may be attributed to bradycardia, low blood pressure, hypothyroidism, or other entities.
  Some patients very often have bradycardia in the ECG taken in the office and normal HR in the 24 Holter monitoring, the opposite is also possible.
  Patients with bradycardia (without medication or physiological condition as exersice affecting heart rate) in at least 2 ECG (less 60 bpm) and at least 2 Holter monitoring will be analyzed,
  Other variables to consider are:
  Age, gender, blood pressure group, adaptability group, maximum HR in the treadmill test, white coat or masked hypertension, Tilt-Table-test result or syncope cause, Electrophysiological study if available.
  The acknowledge of this phenomenon could have clinical implications in the diagnosis of sick sinus syndrome and physiopathological ones.
Reversible Bradycardia Mimicking Sinus Node Dysfunction as a Manifestation of Subacute Autonomic Nervous System Dysfunction (ANSD). | 2 years
  Bradycardia is the classical presentation form for sinus node dysfunction, mainly when associated with symptoms. Chronotropic incompetence is also a manifestation. Absence of medications with effects on the heart rate (HR) must be ruled out.
  Variables
  1. HR at the ECG, Holter monitoring, stress text, and at the physical examination previous to pacemaker implantation,
  2. Electrophysiological study (EPS): Basic cycle length, Sino-atrial conduction time, Sinus node recovery time, Corrected sinus node recovery time, Intrinsic HR when available 3. Pacemaker variables: HR at day and night or rest time Percentage of stimulation in A and V chambers 4. Syncope: Clinical characteriscs and clinical score Tilt table test results Trans Thoracic Echocardiogram in rest and or stress text Hypothesis: patients with ANSD will start to decrease the percentage atrial stimulation.
Description of the blood pressure hemodynamic profile at a medical office and their prognostic implications. | Three years
  A non invasive, beat to beat BP monitoring, with the ability to measure BP, HR, Cardiac Output and Systemic Vascular Resistance (SVR) was started to use in the EHAR registry since May 2017. A description of this variables in the three BP groups will be collected in the data base (DB).
  This will allow to characterize whether SVR and/or CO maintain BP. Until now BP levels are related with prognosis. In the prognosis model SVR and CO will be add them to know what matter the most: BP levels, SVR and/or CO? In the EHAR registry a collection of the variables recognized as a risk factor for several comorbidities are available to adjust in multivariable analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Eduardo Medina, MD., Principal Investigator — Researcher
Locations (1):
- CES University, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Medina E, Uribe W, Duque M, Alzate L. Past Medical History in patients with Orthostatic Intolerance. XIth International Symposium on the Autonomic Nervous System, Puerto Rico, 24-30. October 2000. Clin Auton Res 2000, 10:258. Summary.
- [Background] Medina E, Uribe W, Duque M, Alzate L. Initial Medical Complain and Symptoms in Patients with Orthostatic Intolerance. XIth International symposium on the autonomic nervous system, Puerto Rico, 24-30 October 2000. Clin Auton Res 2000, 10:258. Summary
- [Background] Medina E, Uribe W, Duque M, Alzate L. Syncope characterization in patients with orthostatic intolerance. XIth International symposium on the autonomic nervous system, Puerto Rico, 24-30 October 2000. Clin Auton Res 2000, 10:243. Summary.
- [Background] Medina E, Uribe W, Duque M, Alzate L. Patients with orthostatic Intolerance: are those with syncope different from those without? Is syncope an acceptable endpoint for therapy? XIth International Symposium on the Autonomic Nervous System, Puerto Rico, 24-30 October 2000. Clin Auton Res 2000, 10:243. Summary
- [Background] Medina E, Uribe W, Duque M, Alzate L. Variation of arterial blood pressure and heart rate during follow up in patients with orthostatic intolerance. XIth International symposium on the autonomic nervous system, Puerto Rico, 24-30 October 2000. Summary.
- [Background] Medina E, Uribe W, Duque M, Alzate L. Severity of Compromise and level of Limitation in patients with Orthostatic Intolerance. XIth International Symposium on the autonomic nervous system, Puerto Rico, 24-30 October 2000. Summary
- [Background] Medina E, Uribe W, Duque M, Alzate L. Diagnosis of orthostatic intolerance based on blood pressure and heart rate characterization. Could symptoms be enough?. XIth International symposium on the autonomic nervous system, Puerto Rico, 24-30 October 2000. Summary
- [Background] Medina L, Mármol A, Duque M, Ossaba S, Uribe W, Olaya M, Marín J, Torres Y, Velásquez J. The tilt table test protocol: How can be improved? Clinical Autonomic Research. Vol 14, Number 5, 2004, page. 310. October 2000. Summary
- [Background] Medina L, Olaya M, Duque M, Restrepo F, Uribe W, Marín J, Velásquez J, Torres Y. Fatigue: a clue symptom in chronic orthostatic disorder. How can it be explained? Clinical Autonomic Research. Vol 14, Number 5, 2004, page. 310. October 2000. Summar
- [Background] L Medina, W Uribe, M Duque, I Melguizo, JM Cotes, Y Torres, MA Restrepo, J Marín, E Gil, J Velasquez. Cardiology and autonomic nervous system department. Clínica Medellín, Universidad CES, Universidad Nacional. Medellín, Colombia. Personality type: a variable associated with biological measures in patients with orthostatic intolerance. 16th International symposium on the autonomic nervous system. Los Cabos, Mexico. October 6-9 2005. Clinical Autonomic Research. Vol 15, number 5, page 346, 2005. Summary.
- [Background] L Medina, W Uribe, M Duque, I Melguizo, JM Cotes, Y Torres, MA Restrepo, J Marín, E Gil, J Velasquez. Cardiology and autonomic nervous system department. Clínica Medellín, Universidad CES, Universidad Nacional. Medellín, Colombia. Descriptive analysis and confidence limits at 95% of stress, depression, SF36, and tilt-test variables in an orthostatic intolerant population. 16th International symposium on the autonomic nervous system. Los Cabos, Mexico, October 6-9 2005. Clinical Autonomic Research. Vol 15, number 5, page 342, 2005. Summary.
- [Background] L Medina, D Aristizabal, M Duque, W Uribe, I Melguizo, JM Cotes, Y Torres, MA Restrepo, J Marín, E Gil, J Velásquez, BLF Restrepo. Cardiology and autonomic nervous system department. Clínica Medellín, Universidad CES, Universidad Nacional and Universidad de Antioquia. Medellín, Colombia. Insulin and glucose metabolism in patients with orthostatic intolerance. 16th International symposium on the autonomic nervous system. Los Cabos, Mexico. October 6-9 2005. Clinical Autonomic Research. Vol 15, number 5, page 333, 2005. Summary.
- [Background] L Medina, M Duque, E Gil, JM Cotes, Marín J, D Bravo, E Gonzalez, MA Restrepo, D Aristizabal, Y Torres, M Jimenez, W Uribe. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Applying tilt testing to diagnose sick sinus syndrome: Does it play role beyond syncope? 17th International symposium on the autonomic nervous system. Westin Riomar, Rio Grande, Puerto Rico, November 1-4 2006. Clinical Autonomic Research. Vol 16, number 5, page 349, 2006. Summary.
- [Background] L Medina , J McEween, J Mendez, W Uribe, M Duque, Marín J E Gil, D Bravo, E Gonzalez, MA Restrepo, Torres Y, Cotes JM. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Hemodynamic effects of the 16 Gly/Arg polymorphism at the ADRB2 gene in hypotensive and hypertensive patients. 17th International symposium on the autonomic nervous system. Westin Riomar, Rio Grande, Puerto Rico, November 1-4 2006. Clinical Autonomic Research. Vol 16, Number 5, page 333, 2006. Summary.
- [Background] L Medina, D Aristizabal, J McEween, J Mendez, W Uribe, Duque M, Marín J E Gil, D Bravo, E Gonzalez, MA Restrepo, Torres Y, Cotes JM. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Diagnostic impact of the syncope symptom score in structurally normal hearts in patients undergoing tilt table testing. 17th International Symposium on the Autonomic Nervous System. Westin Riomar, Rio Grande, Puerto Rico, November 1-4 2006. Clinical Autonomic Research. Vol 16, Number 5, page 342, 2006. Summary.
- [Background] LE Medina, D Aristizabal, J Gallo, J Ochoa, Y Torres, L Montoya, M Correa, R Restrepo, D Moreno, MO Correa, N Zapata, PA Gil, M Franco. Medellin heart study. Study design and distribution by blood pressure, including hypotension. Clinical Autonomic Research. Vol 18, Number 5, page 277, 2008. (Summary).
- [Background] Medina L, Duque M, Marin J, Gonzalez E, Astudillo V, Aristizabal J, Bernal J, Restrepo MA, Arroyave A, Jaramillo G, Torres Y, Uribe W. Essential hypotension registry: Sympathovagal balance at 24 hours, day and night in ambulatory Holter monitoring according to blood pressure groups in real-life settings. Clinical Autonomic Research. Vol 19, Number 5, page 300, 2009. Summary.
- [Background] Medina LE, Duque M, Uribe W, Aristizabal J, Velasquez J, Restrepo MA, Miranda A, Torres Y, Marin J. The essential hypotension registry. Blood pressure at the office and at 24 h ambulatory monitoring is different between groups of essential hypertension, normotension and essential hypotension. Clinical Autonomic Research. Vol 20, number 2, page 139, 2010. Summary.
- [Background] Medina LE, Marin J, Duque M, Uribe W, Mesa S, Aristizabal J, Velasquez J, Restrepo MA, Miranda A, Bernal J, Torres Y. Vasovagal syncope and their relationship with hypotension: What is the current conception and how it may change if essential hypotensive population emerges. The essential hypotension registry. Clinical Autonomic Research. Vol 21, number 2, page 127, 201. Summary
- [Background] Medina L, Duque M, Marin J, Gonzalez E, Astudillo V, Aristizabal J, Bernal J, Restrepo MA, Arroyave A, Jaramillo G, Torres Y, Uribe W. Syncope diagnosis in patients with not apparent structurally heart disease and components for both: neurally mediated and cardiac origin (mixed syncope): is it a quantitative history score reliable? Clinical Autonomic Research. Vol 19, number 5, page 308, 2009. Summary.
- [Background] Medina L. Essential hypotension registry. Cardiovascular Reactivity: A search for the integration of the neuro-cardiovascular relationship and their association with glucose challenge and depression. Clinical Autonomic Research. Vol 19, number 5, page 300, 2009. Summary
- [Background] LE Medina, Aristizabal D, McEween J, W Uribe, Duque M, Marín J Gil E, Bravo D, Gonzalez E, Restrepo MA, Torres Y, Cotes JM. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Are there insulin sensitivity differences expected along the blood pressure spectrum? 17th International symposium on the autonomic nervous system. Westin Riomar, Rio Grande, Puerto Rico, November 1-4 2006. Clinical Autonomic Research. Vol 16, number 5, page 332, 2006. Summary
- [Background] LE Medina, W Uribe, M Duque, E Gonzalez, G Montero, D Bravo, MA Restrepo, M Jimenez, D Aristizábal, T Torres, J Marín. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Does essential or primary hypotension matter? Second joint meeting of the European Federation of Autonomic Societies and the American Autonomic Society. Palais Ferstel. Vienna, Austria. October 10-13, 2007. Clinical Autonomic Research. Vol 17, number 5, page 304, 2007. Summary.
- [Background] LE Medina, J Marín, W Uribe, M Duque, E Gonzalez, G Montero, D Bravo, MA Restrepo, M Jimenez, D Aristizabal. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Population characterization according to blood pressure. Are essential hypotensive different from other blood pressure groups? Second joint meeting of the European Federation of Autonomic Societies and the American Autonomic Society. Palais Ferstel. Vienna, Austria. October 10-13, 2007. Clinical Autonomic Research. Vol 17, number 5, page 304, 2007. Summary
- [Background] LE Medina, W Uribe, J Marín, E Gonzalez, G Montero, D Bravo, MA Restrepo, M Jimenez, D Aristizabal, M Duque. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. The importance of arterial hypotension in the chronic fatigue syndrome. Second joint meeting of the European Federation of Autonomic Societies and the American Autonomic Society. Palais Ferstel. Vienna, Austria. October 10-13, 2007. Clinical Autonomic Research. Vol 17, number 5, page 318, 2007. Summary.
- [Background] LE Medina, M Duque, J Marín, E Gonzalez, G Montero, D Bravo, MA Restrepo, M Jimenez, D Aristizabal, W Uribe. Cardiology and autonomic nervous system department. Clínica Medellín, Medellín, Colombia. Are there differences in the variables hemoglobin, hematocrit and ferritin between normotensive patients and essential hypertensive and hypotensive? Second joint meeting of the European Federation of Autonomic Societies and the American Autonomic Society. Palais Ferstel. Vienna, Austria. October 10-13, 2007. Clinical Autonomic Research. Vol 17, number 5, page 311, 2007. Summary
- [Background] LE Medina, J Ospina, MA Lemos, G Cuartas, D Aristizabal, J Calle, Gutierrez, Y Torres. Relationship between blood pressure, depression and anxiety. A step into the concept of psychobiotype (mind-body relationship). Clinical Autonomic Research. Vol 18, number 5, page 277, 2008. Summary
- [Background] LE Medina, W Uribe, J Marin, G Montero, B Astudillo, MA Restrepo, J Bernal, Y Torres, M Duque. Blood pressure characterization in essentials hypotension and/or orthostatic hypotension. Clinical Autonomic Research. Vol 18, number 5, page 277, 2008. Summary.
- [Background] Medina L, Uribe W, Marin J, Gonzalez E, Astudillo V, Aristizabal J, Velasquez J, Bernal J, Torres Y, Duque M. Chronotropic incompetence in the head-up tilt testing: a useful diagnostic marker or clinically irrelevant finding? Accepted for publication at the European Heart Journal, 2009 (Summary).
- [Background] Medina L. Essential Hypotension registry: Definition, blood pressure and demographic report. Clinical Autonomic Research. Vol 19, number 5, page 308, 2009. Summary
- [Background] Medina LE, Ospina J, Lemos MA, Cuartas G, Calle J, Gutierrez M, Torres Y. Essential hypotension registry: Psychometric measurements for anxiety, depression and coping strategies: Hypotension is associated with depression and anxiety. Is there a psycho-biotype? Preliminary Report. Clinical Autonomic Research. Vol 19, number 5, page 296, 2009. Summary
- [Background] Medina LE, Duque M, Uribe W, Aristizabal J, Velasquez J, Restrepo MA, Miranda A, Torres Y, Marin J. It is glucose metabolism (HOMA and the relation: 2 h postprandial plasma glucose/fasting glucose) different between blood pressure groups? The essential hypotension registry. Clinical Autonomic Research. Vol 20, number 2, page 139, 2010. Summary.
- [Background] Medina LE, Duque M, Marin J, Aristizabal J, Velasquez J, Miranda A, Torres Y, Restrepo MA, Uribe W. The essential hypotension registry. Rationale for the blood pressure classification and the importance of the stress response. Clinical Autonomic Research. Vol 20, number 2, page 139, 2010. Summary
- [Background] Medina LE, Uribe W, Marin J, Aristizabal J, Velasquez J, Miranda A, Torres Y, Restrepo MA, Duque M. What do patients with classical and initial orthostatic hypotension, without an identifiable cause have to teach us? The essential hypotension registry. Description of the population and the blood pressure measurements. Clinical Autonomic Research. Vol 20, number 2, page 140, 2010. Summary
- [Background] Medina LE, Uribe W, Marin J, Aristizabal J, Velasquez J, Miranda A, Torres Y, Restrepo MA, Duque M. The importance of essential hypotension in syncope. A report of 877 patients. The essential hypotension registry. Clinical. Autonomic Research. Vol 20, number 2, page 140, 2010. Summary
- [Background] Huber M, Knottnerus JA, Green L, van der Horst H, Jadad AR, Kromhout D, Leonard B, Lorig K, Loureiro MI, van der Meer JW, Schnabel P, Smith R, van Weel C, Smid H. How should we define health? BMJ. 2011 Jul 26;343:d4163. doi: 10.1136/bmj.d4163. No abstract available. PMID 21791490
- [Background] Godly F. What is health? BMJ 2011; 343: d4817
- [Background] Pacak K, Palkovits M. Stressor specificity of central neuroendocrine responses: implications for stress-related disorders. Endocr Rev. 2001 Aug;22(4):502-48. doi: 10.1210/edrv.22.4.0436. PMID 11493581
- [Background] Accurso V, Winnicki M, Shamsuzzaman AS, Wenzel A, Johnson AK, Somers VK. Predisposition to vasovagal syncope in subjects with blood/injury phobia. Circulation. 2001 Aug 21;104(8):903-7. doi: 10.1161/hc3301.094910. PMID 11514377
- [Background] Karatsoreos IN, McEwen BS. Resilience and vulnerability: a neurobiological perspective. F1000Prime Rep. 2013 May 1;5:13. doi: 10.12703/P5-13. Print 2013. PMID 23710327
- [Background] Bernard, Claude. Le phénoménes de la Vie. Paris, 1878.
- [Background] Walter B Cannon, Organization for physiological homeostasis. Physiological Reviews 1929; Vol IX, No 3, 399-430.
- [Background] Walter B Cannon, The Wisdom of the body. Preface and Introduction, page xiii and page 19; 1939, New York: W. M. Norton & Co
- [Background] Selye H. A syndrome produced by diverse nocuous agents. 1936. J Neuropsychiatry Clin Neurosci. 1998 Spring;10(2):230-1. doi: 10.1176/jnp.10.2.230a. No abstract available. PMID 9722327
- [Background] SELYE H. THE STRESS OF LIFE--NEW FOCAL POINT FOR UNDERSTANDING ACCIDENTS. Nurs Forum. 1965;4:28-38. doi: 10.1111/j.1744-6198.1965.tb01011.x. No abstract available. PMID 14280643
- [Background] Ray O. The revolutionary health science of psychoendoneuroimmunology: a new paradigm for understanding health and treating illness. Ann N Y Acad Sci. 2004 Dec;1032:35-51. doi: 10.1196/annals.1314.004. PMID 15677394
- [Background] McEwen BS. Protective and damaging effects of stress mediators. N Engl J Med. 1998 Jan 15;338(3):171-9. doi: 10.1056/NEJM199801153380307. No abstract available. PMID 9428819
- [Background] Rocci R. Un Nuovo Sphigmomanometro. Gazeta Medica Di Torino.1896; 50. December 10
- [Background] Korotkoff, NC. On the question of methods of determining the blood pressure. Reports of the Imperial Military Academy, St. Petersburg, 1905; 11: 365
- [Background] Cook, Henry W. Blood Pressure in Prognosis. Med Record, 1911; 80: 959-967.
- [Background] Chrousos GP. The hypothalamic-pituitary-adrenal axis and immune-mediated inflammation. N Engl J Med. 1995 May 18;332(20):1351-62. doi: 10.1056/NEJM199505183322008. No abstract available. PMID 7715646
- [Background] Gruzelier J, Clow A, Evans P, Lazar I, Walker L. Mind-body influences on immunity: lateralized control, stress, individual differences predictors, and prophylaxis. Ann N Y Acad Sci. 1998 Jun 30;851:487-94. doi: 10.1111/j.1749-6632.1998.tb09027.x. No abstract available. PMID 9668642
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186
- [Background] Shin C, Abbott RD, Lee H, Kim J, Kimm K. Prevalence and correlates of orthostatic hypotension in middle-aged men and women in Korea: the Korean Health and Genome Study. J Hum Hypertens. 2004 Oct;18(10):717-23. doi: 10.1038/sj.jhh.1001732. PMID 15116144
- [Background] Fedorowski A, Stavenow L, Hedblad B, Berglund G, Nilsson PM, Melander O. Orthostatic hypotension predicts all-cause mortality and coronary events in middle-aged individuals (The Malmo Preventive Project). Eur Heart J. 2010 Jan;31(1):85-91. doi: 10.1093/eurheartj/ehp329. Epub 2009 Aug 20. PMID 19696189
- [Background] Rose KM, Eigenbrodt ML, Biga RL, Couper DJ, Light KC, Sharrett AR, Heiss G. Orthostatic hypotension predicts mortality in middle-aged adults: the Atherosclerosis Risk In Communities (ARIC) Study. Circulation. 2006 Aug 15;114(7):630-6. doi: 10.1161/CIRCULATIONAHA.105.598722. Epub 2006 Aug 7. PMID 16894039
- [Background] Rose KM, Tyroler HA, Nardo CJ, Arnett DK, Light KC, Rosamond W, Sharrett AR, Szklo M. Orthostatic hypotension and the incidence of coronary heart disease: the Atherosclerosis Risk in Communities study. Am J Hypertens. 2000 Jun;13(6 Pt 1):571-8. doi: 10.1016/s0895-7061(99)00257-5. PMID 10912737
- [Background] Benvenuto LJ, Krakoff LR. Morbidity and mortality of orthostatic hypotension: implications for management of cardiovascular disease. Am J Hypertens. 2011 Feb;24(2):135-44. doi: 10.1038/ajh.2010.146. Epub 2010 Sep 2. PMID 20814408
- [Background] The Autonomic Nervous System in Health and Disease. Edited by David S. Goldstein. Marcel Dekker editors, New York, 2001, pages 480-490.
- [Background] Ferrier C, Esler MD, Eisenhofer G, Wallin BG, Horne M, Cox HS, Lambert G, Jennings GL. Increased norepinephrine spillover into the jugular veins in essential hypertension. Hypertension. 1992 Jan;19(1):62-9. doi: 10.1161/01.hyp.19.1.62. PMID 1730441
- [Background] Staessen J, Amery A, Fagard R. Isolated systolic hypertension in the elderly. J Hypertens. 1990 May;8(5):393-405. doi: 10.1097/00004872-199005000-00001. No abstract available. PMID 2163412
- [Background] Kannel WB, Wolf PA, McGee DL, Dawber TR, McNamara P, Castelli WP. Systolic blood pressure, arterial rigidity, and risk of stroke. The Framingham study. JAMA. 1981 Mar 27;245(12):1225-9. PMID 7206111
- [Background] Miall WE. Systolic or diastolic hypertension--which matters most? Clin Exp Hypertens A. 1982;4(7):1121-31. doi: 10.3109/10641968209060779. PMID 7116661
- [Background] Miall WE, Lovell HG. Relation between change of blood pressure and age. Br Med J. 1967 Jun 10;2(5553):660-4. doi: 10.1136/bmj.2.5553.660. No abstract available. PMID 6024522
- [Background] Grassi G. Assessment of sympathetic cardiovascular drive in human hypertension: achievements and perspectives. Hypertension. 2009 Oct;54(4):690-7. doi: 10.1161/HYPERTENSIONAHA.108.119883. Epub 2009 Aug 31. PMID 19720958
- [Background] Franklin SS, Gustin W 4th, Wong ND, Larson MG, Weber MA, Kannel WB, Levy D. Hemodynamic patterns of age-related changes in blood pressure. The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):308-15. doi: 10.1161/01.cir.96.1.308. PMID 9236450
- [Background] Acelajado M, Calhoun D, Oparil S. Pathogenesis of hypertension. In: Hypertension. A Companion of Branwalds heart disease, 2nd Edition, 2013, Chapter 2, page 12, Elsevier Saunders, Philadelphia
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Background] Pickering TG, Shimbo D, Haas D. Ambulatory blood-pressure monitoring. N Engl J Med. 2006 Jun 1;354(22):2368-74. doi: 10.1056/NEJMra060433. No abstract available. PMID 16738273
- [Background] Kikuya M, Hansen TW, Thijs L, Bjorklund-Bodegard K, Kuznetsova T, Ohkubo T, Richart T, Torp-Pedersen C, Lind L, Ibsen H, Imai Y, Staessen JA; International Database on Ambulatory blood pressure monitoring in relation to Cardiovascular Outcomes Investigators. Diagnostic thresholds for ambulatory blood pressure monitoring based on 10-year cardiovascular risk. Circulation. 2007 Apr 24;115(16):2145-52. doi: 10.1161/CIRCULATIONAHA.106.662254. Epub 2007 Apr 9. PMID 17420350
- [Background] Beckett NS, Peters R, Fletcher AE, Staessen JA, Liu L, Dumitrascu D, Stoyanovsky V, Antikainen RL, Nikitin Y, Anderson C, Belhani A, Forette F, Rajkumar C, Thijs L, Banya W, Bulpitt CJ; HYVET Study Group. Treatment of hypertension in patients 80 years of age or older. N Engl J Med. 2008 May 1;358(18):1887-98. doi: 10.1056/NEJMoa0801369. Epub 2008 Mar 31. PMID 18378519
- [Background] Diseases and Conditions Index - Hypotension. National Heart Lung and Blood Institute. September 2008.
- [Background] Low blood pressure (hypotension) - Definition. MayoClinic.com. Mayo Foundation for Medical Education and Research. 2009/05/23.
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Robertson D. The pathophysiology and diagnosis of orthostatic hypotension. Clin Auton Res. 2008 Mar;18 Suppl 1:2-7. doi: 10.1007/s10286-007-1004-0. Epub 2008 Mar 27. PMID 18368300
- [Background] Task Force for the Diagnosis and Management of Syncope; European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Heart Failure Association (HFA); Heart Rhythm Society (HRS); Moya A, Sutton R, Ammirati F, Blanc JJ, Brignole M, Dahm JB, Deharo JC, Gajek J, Gjesdal K, Krahn A, Massin M, Pepi M, Pezawas T, Ruiz Granell R, Sarasin F, Ungar A, van Dijk JG, Walma EP, Wieling W. Guidelines for the diagnosis and management of syncope (version 2009). Eur Heart J. 2009 Nov;30(21):2631-71. doi: 10.1093/eurheartj/ehp298. Epub 2009 Aug 27. No abstract available. PMID 19713422
- [Background] Carter JR, Ray CA. Sympathetic neural responses to mental stress: responders, nonresponders and sex differences. Am J Physiol Heart Circ Physiol. 2009 Mar;296(3):H847-53. doi: 10.1152/ajpheart.01234.2008. Epub 2009 Jan 23. PMID 19168718
- [Background] Sheldon R, Rose S, Connolly S, Ritchie D, Koshman ML, Frenneaux M. Diagnostic criteria for vasovagal syncope based on a quantitative history. Eur Heart J. 2006 Feb;27(3):344-50. doi: 10.1093/eurheartj/ehi584. Epub 2005 Oct 13. PMID 16223744
- [Background] Medina LE, Duque M, Uribe W. Initial medical complaints in patients with orthostatic intolerance. Clin Auton Res 2000, 10: 258 (Summary).
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Grubb BP, Kosinski DJ, Boehm K, Kip K. The postural orthostatic tachycardia syndrome: a neurocardiogenic variant identified during head-up tilt table testing. Pacing Clin Electrophysiol. 1997 Sep;20(9 Pt 1):2205-12. doi: 10.1111/j.1540-8159.1997.tb04238.x. PMID 9309745
- [Background] Bybee KA, Kara T, Prasad A, Lerman A, Barsness GW, Wright RS, Rihal CS. Systematic review: transient left ventricular apical ballooning: a syndrome that mimics ST-segment elevation myocardial infarction. Ann Intern Med. 2004 Dec 7;141(11):858-65. doi: 10.7326/0003-4819-141-11-200412070-00010. PMID 15583228
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Raiha I, Luutonen S, Piha J, Seppanen A, Toikka T, Sourander L. Prevalence, predisposing factors, and prognostic importance of postural hypotension. Arch Intern Med. 1995 May 8;155(9):930-5. doi: 10.1001/archinte.1995.00430090067008. PMID 7726701
- [Background] Furlan R, Jacob G, Palazzolo L, Rimoldi A, Diedrich A, Harris PA, Porta A, Malliani A, Mosqueda-Garcia R, Robertson D. Sequential modulation of cardiac autonomic control induced by cardiopulmonary and arterial baroreflex mechanisms. Circulation. 2001 Dec 11;104(24):2932-7. doi: 10.1161/hc4901.100360. PMID 11739308
- [Background] White W, Shah H. Ambulatory blood pressure monitoring in clinical hypertension management. In: Hypertension. A Companion to Branwald Heart Disease, 2013, Second edition, Chapter 6, Page 59. Edited by Black H and Elliot W.
- [Background] Devereux RB, Reichek N. Echocardiographic determination of left ventricular mass in man. Anatomic validation of the method. Circulation. 1977 Apr;55(4):613-8. doi: 10.1161/01.cir.55.4.613. PMID 138494
- [Background] Patel MR, Bailey SR, Bonow RO, Chambers CE, Chan PS, Dehmer GJ, Kirtane AJ, Wann LS, Ward RP. ACCF/SCAI/AATS/AHA/ASE/ASNC/HFSA/HRS/SCCM/SCCT/SCMR/STS 2012 appropriate use criteria for diagnostic catheterization: a report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, Society for Cardiovascular Angiography and Interventions, American Association for Thoracic Surgery, American Heart Association, American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Failure Society of America, Heart Rhythm Society, Society of Critical Care Medicine, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2012 May 29;59(22):1995-2027. doi: 10.1016/j.jacc.2012.03.003. Epub 2012 May 9. PMID 22578925
- [Background] Electrophysiological testing, Chapter 4, page 62. In: Clinical Arhythmology and Electrophysiology. A Companion of Branwald´s Heart Disease, 2nd Ed. Elsevir, Saunders 2012; Philadelphia. Edited by Ziad F. Issa, John M Miller, Douglas P. Zipes
- [Background] Narula OS, Samet P, Javier RP. Significance of the sinus-node recovery time. Circulation. 1972 Jan;45(1):140-58. doi: 10.1161/01.cir.45.1.140. No abstract available. PMID 4108657
- [Background] Chadda KD, Banka VS, Bodenheimer MM, Helfant RH. Corrected sinus node recovery time. Experimental physiologic and pathologic determinants. Circulation. 1975 May;51(5):797-801. doi: 10.1161/01.cir.51.5.797. PMID 1122582
- [Background] Issa Z, Miller J, Zipes D. Sinus Node Dysfunction. In: Clinical arrhythmology and electrophysiology. A Companion to Branwald Heart Disease, 2012, Second edition, Chapter 8, Page 164. Edited by Issa Z, Miller J, Zipes D.
- [Background] Desai JM, Scheinman MM, Strauss HC, Massie B, O'Young J. Electrophysiologic effects on combined autonomic blockade in patients with sinus node disease. Circulation. 1981 Apr;63(4):953-60. doi: 10.1161/01.cir.63.4.953. PMID 7471352
- [Background] Medina L, Uribe W, Marin J, Gonzalez E, Astudillo V, Aristizabal J, Velasquez J, Bernal J, Torres Y, Duque M. Chronotropic incompetence in the head-up tilt testing: a useful diagnostic marker or clinically irrelevant finding? European Heart Journal, 2009 (Summary).
- [Background] Inappropriate Sinus Tachycardia, Chapter 16, page 375. In: Clinical Arhythmology and Electrophysiology. A Companion of Branwald´s Heart Disease, 2nd Ed. Elsevir, Saunders 2012; Philadelphia. Edited by Ziad F. Issa, John M Miller, Douglas P. Zipes.
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Zivin J. Ischemic cerebrovascular disease. In: Cecil Medicine 24th Edition, Edited by Goldman Lee and Schafer A. 2012, Elsevier Sanders, Inc. Philadelphia. Page 2304, Chapter 413.
- [Background] Albers GW, Caplan LR, Easton JD, Fayad PB, Mohr JP, Saver JL, Sherman DG; TIA Working Group. Transient ischemic attack--proposal for a new definition. N Engl J Med. 2002 Nov 21;347(21):1713-6. doi: 10.1056/NEJMsb020987. No abstract available. PMID 12444191
- [Background] Inzucchi S, Sherwin R. Type II Diabetes Mellitus. In: Cecil Medicine 24th Edition, Edited by Goldman Lee and Schafer A. 2012, Elsevier Sanders, Inc. Philadelphia. Page 1690, Chapter 237.
- [Background] Fukuda K, Straus SE, Hickie I, Sharpe MC, Dobbins JG, Komaroff A. The chronic fatigue syndrome: a comprehensive approach to its definition and study. International Chronic Fatigue Syndrome Study Group. Ann Intern Med. 1994 Dec 15;121(12):953-9. doi: 10.7326/0003-4819-121-12-199412150-00009. PMID 7978722
- [Background] Andersen MM, Permin H, Albrecht F. Illness and disability in Danish Chronic Fatigue Syndrome patients at diagnosis and 5-year follow-up. J Psychosom Res. 2004 Feb;56(2):217-29. doi: 10.1016/S0022-3999(03)00065-5. PMID 15016582
- [Background] Bennett R. Fibromyalgia, chronic fatigue syndrome, and myofascial pain. Curr Opin Rheumatol. 1998 Mar;10(2):95-103. doi: 10.1097/00002281-199803000-00002. PMID 9567202
- [Background] McEwen BS, Gianaros PJ. Central role of the brain in stress and adaptation: links to socioeconomic status, health, and disease. Ann N Y Acad Sci. 2010 Feb;1186:190-222. doi: 10.1111/j.1749-6632.2009.05331.x. PMID 20201874
- [Background] Andersson U, Tracey KJ. Reflex principles of immunological homeostasis. Annu Rev Immunol. 2012;30:313-35. doi: 10.1146/annurev-immunol-020711-075015. Epub 2012 Jan 6. PMID 22224768
- [Background] Parati G, Stergiou G, O'Brien E, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. European Society of Hypertension practice guidelines for ambulatory blood pressure monitoring. J Hypertens. 2014 Jul;32(7):1359-66. doi: 10.1097/HJH.0000000000000221. PMID 24886823